CLINICAL TRIAL: NCT02403193
Title: Phase I/Ib Trial of Single Agent PBF-509 and in Combination With PDR001 for Patients With Advanced NSCLC
Brief Title: Trial of PBF-509 and PDR001 in Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Acronym: AdenONCO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Palobiofarma SL (Industry)
Collaborators: Novartis (Industry); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC18321
Record Dates: First submitted 2015-03-17; First posted 2015-03-31 (Estimated); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Adenosine A2a receptor antagonist; NSCLC; PBF-509; Immunotherapy; adenosine; PDR001; immune checkpoint inhibitors; Programmed Death-1 (PD-1) receptor; Adenosine A2a receptor (A2AR)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- PBF-509_80 mg (Experimental)
  Interventions: Drug: PBF-509_80 mg
- PBF-509_160 mg (Experimental)
  Interventions: Drug: PBF-509_160 mg
- PBF-509_320 mg (Experimental)
  Interventions: Drug: PBF-509_320 mg
- PBF-509_640 mg (Experimental)
  Interventions: Drug: PBF-509_640 mg
- PBF509_160 mg +PDR001 (Experimental)
  Interventions: Drug: Combo PBF-509 (160 mg) + PDR001
- PBF509_320 mg+PDR001 (Experimental)
  Interventions: Drug: Combo PBF-509 (320 mg) + PDR001
- PBF509_640 mg +PDR001 (Experimental)
  Interventions: Drug: Combo PBF-509 (640 mg) + PDR001
- RP2D (PBF-509+PDR001)_immuno naïve (Experimental): Immunotherapy naïve patients will be treated at the combination RP2D previously determined in the phase Ib, dose escalation portion of the trial.
  Interventions: Drug: RP2D (PBF-509+PDR001)_immuno naïve
- RP2D (PBF-509+PDR001)_immuno treated (Experimental): Patients previously treated with immunotherapy (previous immune checkpoint inhibitors; anti-CTLA-4, anti-PD-1, anti-PD-L1 and/or combinations) will be treated at the combination RP2D previously determined in the phase Ib, dose escalation portion of the trial.
  Interventions: Drug: Experimental: RP2D (PBF-509+PDR001)_immuno treated

INTERVENTIONS:
Drug: PBF-509_80 mg — PBF-509: 80 mg, PO, twice daily (BID)
  Arms: PBF-509_80 mg
Drug: PBF-509_160 mg — PBF-509: 160 mg, PO, twice daily (BID)
  Arms: PBF-509_160 mg
Drug: PBF-509_320 mg — PBF-509: 320 mg, PO, twice daily (BID)
  Arms: PBF-509_320 mg
Drug: PBF-509_640 mg — PBF-509: 640 mg, PO, twice daily (BID)
  Arms: PBF-509_640 mg
Drug: Combo PBF-509 (160 mg) + PDR001 — Drug 1: PDR001 administered intravenously. Drug 2: PBF-509 administered orally
  Arms: PBF509_160 mg +PDR001
Drug: Combo PBF-509 (320 mg) + PDR001 — Drug 1: PDR001 administered intravenously. Drug 2: PBF-509 administered orally
  Arms: PBF509_320 mg+PDR001
Drug: Combo PBF-509 (640 mg) + PDR001 — Drug 1: PDR001 administered intravenously. Drug 2: PBF-509 administered orally
  Arms: PBF509_640 mg +PDR001
Drug: RP2D (PBF-509+PDR001)_immuno naïve — Drug 1: PDR001 administered intravenously. Drug 2: PBF509 administered orally
  Arms: RP2D (PBF-509+PDR001)_immuno naïve
Drug: Experimental: RP2D (PBF-509+PDR001)_immuno treated — Drug 1: PDR001 administered intravenously. Drug 2: PBF509 administered orally
  Arms: RP2D (PBF-509+PDR001)_immuno treated

SUMMARY:
The purpose of this study is to determine the safety, tolerability, feasibility and preliminary efficacy of the administration of PBF-509 (Adenosine A2a receptor antagonist) as single agent or in combination with PDR001 (programmed cell death 1 receptor antibody (PD-1 Ab)) to NSCLC patients.

DETAILED DESCRIPTION:
A single institution phase I/Ib (dose escalation plus expansion) clinical trial of PBF-509 and combination treatment of PDR001 plus PBF-509 in Eastern Cooperative Oncology Group (ECOG) 0-1 patients with immunotherapy naïve and pretreated, advanced or metastatic NSCLC will be conducted to evaluate the safety, tolerability and preliminary efficacy of the combination.

The main objectives of the proposed Phase I trial will be:

Phase I Dose Escalation:

* To determine the safety and tolerability of PBF-509 during a phase I dose escalation trial
* Determine the pharmacokinetic profile of PBF-509
* Determine the safety profile of PBF-509

Phase 1 Dose Expansion:

• To further determine safety and tolerability of PBF-509 at the recommended phase II dose (RP2D)

Phase Ib Dose Escalation:

* To determine the dose limiting toxicities (DLT), maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of PBF-509 in combination with PDR001
* To determine the pharmacokinetics (PK) of PBF-509 in combination with PDR001

Phase Ib Expansion:

* To determine the safety and tolerability of PBF-509 in combination with PDR001, at the RP2D, in both immunotherapy naïve and pretreated advanced NSCLC
* To evaluate the response rate (ORR) of PBF-509 in combination with PDR001, at the RP2D, in both immunotherapy naïve and pretreated advanced NSCLC
* To evaluate the progression free (PFS) and overall survival (OS) of PBF-509 in combination with PDR001, at the RP2D, in both immunotherapy naïve and pretreated advanced NSCLC
* To determine the pharmacokinetics (PK) of PBF-509 in combination with PDR001

Correlative (Exploratory) Studies:

* To evaluate the biological activity of PBF-509 alone and in combination with PDR001 by assessment of potential pharmacodynamic (PD) biomarkers in tumor biopsy specimens of patients with advanced NSCLC
* To determine association of pre- or on-treatment expression of other immune checkpoints genes with resistance to single agent PBF-509 and dual immune inhibitory (PDR001+ PBF-509) treatment.
* Determine the pharmacokinetics of PDR001 in combination with PBF-509

The phase I and phase Ib dose escalations will be conducted utilizing the standard 3+3 dose escalation method. Pharmacokinetic (PK) data will be obtained for PBF-509 and PDR001.

The phase Ib dose expansion will consist of 2 independent groups of immunotherapy naïve and pretreated (previous immune checkpoint inhibitors; anti-CTLA-4, anti-PD-1, anti-PD-L1 and/or combinations) patients. Pharmacodynamic (PD) data will be obtained for potential biomarker analysis with pre-treatment and on-treatment tumor biopsies.

Number of Patients:

Phase I Dose escalation and safety expansion: 15-18 patients will be treated with single agent PBF-509 in escalation and up to 20 patients may be treated at the RP2D as a safety expansion group.

Phase Ib Dose escalation: 15-24 patients will be treated

The specific number of patients enrolled will vary depending on whether additional patients could be required during the escalation period if dose de-escalation cohorts or intermediate doses are enrolled, or when a dose-escalation cohort is expanded.

Phase Ib Dose Expansion: 20 patients per group will be enrolled for a total of 40 patients. Assuming 10-15% eligibility/screen failures, a maximum 50 patients will be enrolled.

Safety Assessments:

The maximun tolerated dose (MTD) evaluation will be based on the dose-limiting toxicity (DLT) Evaluable Population which includes all patients enrolled in the dose-escalation portion of the trial, who receive the protocol-assigned treatment with PDR001 and PBF-509 and complete the safety follow-up through the DLT evaluation period, or experience a DLT during the DLT evaluation period.

The safety evaluation will be based on the treated Population, which includes all patients who receive any dose of investigational product, and will include adverse events (AEs), serious adverse event (SAEs), laboratory evaluations and electrocardiogram (ECG) results.

AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 and described by system organ class and preferred tem using the Medical Dictionary for Regulatory Activities (MedDRA). Clinically relevant Laboratory abnormalities with toxicity grades according to the NCI CTCAE v4.03 will be derived and summarized.

Efficacy Assessments:

The efficacy analysis will be based on the treated Population which includes all patients who receive any dose of either investigational product. The following efficacy endpoints will be analyzed:

1. Objective Response Rate (ORR) is defined as confirmed complete response (CR) or partial response (PR) based on modified Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Disease control rate (DCR) is defined as CR, PR, or stable disease (SD) based on modified RECIST v1.1.
2. Duration of response (DoR) is defined as the duration from the first documentation of Objective response (OR) to the first documented disease progression or death due to any cause, whichever occurs first.
3. Progression-free survival (PFS) will be measured from the start of treatment until the documentation of disease progression or death due to any cause, whichever occurs first.
4. Overall survival (OS) will be determined as the time from the start of treatment with PDR001 and PBF-509 until death due to any cause

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologic or cytologic diagnosis of advanced/metastatic NSCLC. For those with mixed histology, there must be a predominant histology.
2. Patients must previously have received at least one prior line of therapy for their disease
3. EGFR mutation with exon 19 deletion or L858R mutation (Exon 21) or ALK rearrangement positive must have failed prior TKI therapy
4. Able, willing to give written consent for available archival tumor samples (not mandatory) and tumor biopsies before and during protocol therapy (mandatory).
5. Prior immunotherapy is allowed (previous immune checkpoint inhibitors; anti-CTLA-4, anti-PD-1, anti-PD-L1 and/or combinations), except for the patients enrolled to the immunotherapy naïve group of the phase IB dose expansion.
6. Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral computed tomography (CT) scan, Magnetic resonance imaging (MRI), or calipers by clinical exam. See Section 13.
7. Written informed consent and any locally-required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
8. Age > 18 years at time of study entry
9. Eastern Cooperative Oncology Group (ECOG) 0-1
10. Adequate normal organ and marrow function
11. Female patients must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old or no menses for 1 year without an alternative medical cause; OR history of complete hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
12. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use 2 highly effective methods of contraception while taking study treatment and for 90 days after the last dose of study treatment.
13. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Symptomatic and/or untreated Brain Metastases
2. Pregnancy or breast feeding
3. Serious uncontrolled medical disorder or active infection that in the investigator's opinion would impair the patient's ability to receive study treatment.
4. Concurrent use of other anticancer approved or investigational agents is not allowed.
5. Active or prior documented autoimmune disease within the past 2 years. NOTE: Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
6. Prior malignancy in past 2 years or as identified in Section 7.2 of this protocol
7. Patients receiving systemic steroids ≥ 10mg/day of prednisone or the equivalent
8. Smoking (cigarettes, cigars or pipes) must be discontinued at least 7 days prior to initiating study drug administration; smoking cessation products (transdermal nicotine patches or chewing gum may be used)
9. Concurrent administration of strong inhibitors or moderate inducers of CYP1A2 is not permitted; administration must be discontinued at least 7 days prior to initiating study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-10; Primary Completion 2021-10 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of PBF-509 as single agent | 28 days
  The MTD evaluation will be based on the DLT Evaluable Population which includes all patients enrolled in the dose-escalation portion of the trial, who receive the protocol-assigned treatment with PBF-509 and complete the safety follow-up through the DLT evaluation period, or experience a DLT during the DLT evaluation period.
Maximum Tolerated Dose (MTD) of the combination (PBF-509+PDR001) treatment | 56 days
  The MTD evaluation will be based on the DLT Evaluable Population which includes all patients enrolled in the dose-escalation portion of the trial, who receive the protocol-assigned treatment with PDR001 and PBF-509 and complete the safety follow-up through the DLT evaluation period, or experience a DLT during the DLT evaluation period.

SECONDARY OUTCOMES:
Time to PBF-509 peak concentration in plasma "Tmax" | 8 days
  The parameter will be calculated from plasma samples collected at days 1 and 8 after drug administration.
  It will consist in the time (in minutes) to reach the maximum "PBF-509" concentration in plasma samples of patients after oral administration of PBF-509.
Time to PBF-509 peak concentration in plasma at steady state "Tmax,ss" | 8 days
  The parameter will be calculated from plasma samples collected at days 1 and 8 after drug administration.
  It will consist in the time (in minutes) to reach the maximum "PBF-509" concentration in plasma samples of patients during a dosing interval at steady state.
PBF-509 peak concentration in plasma "Cmax" | 8 days
  The parameter will be calculated from plasma samples collected at days 1 and 8 after drug administration.
  It will consist in the maximum plasma concentration (ng/mL) of PBF-509 observed after administration.
PBF-509 peak concentration in plasma at steady state"Cmax,ss" | 8 days
  The parameter will be calculated from plasma samples collected at days 1 and 8 after drug administration.
  It will consist in the maximum plasma concentration (ng/mL) of PBF-509 observed during a dosing interval at steady state.
The area under PBF-509 plasma concentration-time curve to infinite time "AUC(0-inf)" | 8 days
  The parameter will be calculated from plasma samples collected at days 1 and 8 after drug administration.
  It will consist in the area under the concentration-time curve from zero up to ∞ with extrapolation of the terminal phase. "AUC(0-inf)" will be given in Amount·time/ volume units
The area under PBF-509 plasma concentration-time curve up to time 't' "AUC(0-t)" | 8 days
  The parameter will be calculated from plasma samples collected at days 1 and 8 after drug administration.
  It will consist in the area under the concentration-time curve from zero up to a definite time t. "AUC(0-t)" will be given in Amount·time/ volume units.
The area under PBF-509 plasma concentration-time curve over the dosing interval "AUC(0-τ)" | 8 days
  The parameter will be calculated from plasma samples collected at days 1 and 8 after drug administration.
  It will consist in the area under the concentration-time curve over the dosing interval. "AUC(0-τ)" will be given in Amount·time/ volume units.
PBF-509 half-life in plasma " t½" | 8 days
  The parameter will be calculated from plasma samples collected at days 1 and 8 after drug administration.
  It will consist in the terminal half-life of PBF-509 in plasma. "t½" will be given in hours (h)
PBF-509 apparent volume of distribution following extravascular administration"Vd/F" | 8 days
  The parameter will be calculated from plasma samples collected at days 1 and 8 after drug administration.
  It will consist in the apparent volume of distribution during terminal phase after oral / extravascular administration. "Vd/F" will be given in Volume or volume/kg units.
PBF-509 total body clearance following extravascular administration "Cl/F" | 8 days
  The parameter will be calculated from plasma samples collected at days 1 and 8 after drug administration.
  It will consist in the apparent total plasma or serum clearance of drug after oral administration. "Cl/F" will be given in the Volume/ time or volume/ time/ kg units.
The PBF 509 accumulation index "Rac" | 8 days
  The parameter will be calculated from plasma samples collected at days 1 and 8 after drug administration.
  It will consist in the accumulation ratio calculated from Cmax,ss at steady state and Cmax after single dosing.
Efficacy as measured by Objective response rate (ORR) | 3 years
  ORR: Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).
  ORR is defined as confirmed complete response (CR) or partial response (PR) based on modified RECIST v1.1.
Efficacy as measured by Disease control rate (DCR) | 3 years
  The disease control rate (DCR) will be estimated considering the following variables:
  Complete response (CR), Partial response (PR) and stable disease (SD) as described by Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).
  These variables will be assessed based on Imaging-based evaluation methods as chest x-ray, conventional computed tomography (CT) and magnetic resonance imaging (MRI) that will be performed every 2 cycles of 28 days administration
Efficacy as measured by duration of response (DoR) | 3 years
  Duration of response (DoR) is defined as the duration from the first documentation of OR to the first documented disease progression or death due to any cause, whichever occurs first.
Efficacy as measured by progression-free survival (PFS) | 3 years
  Progression-free survival (PFS) will be measured from the start of treatment until the documentation of disease progression or death due to any cause, whichever occurs first. For subjects who are alive and progression-free at the time of data cut-off for analysis, PFS will be censored at the last tumor assessment date.
Efficacy as measured by overall survival (OS) | 3 years
  Overall survival (OS) will be determined as the time from the start of treatment until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Chiappori, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- H.Lee Moffitt Cancer center, Tampa, Florida, United States

REFERENCES:
- [Derived] Chiappori AA, Creelan B, Tanvetyanon T, Gray JE, Haura EB, Thapa R, Barlow ML, Chen Z, Chen DT, Beg AA, Boyle TA, Castro J, Morgan L, Morris E, Aregay M, Hurtado FK, Manenti L, Antonia S. Phase I Study of Taminadenant (PBF509/NIR178), an Adenosine 2A Receptor Antagonist, with or without Spartalizumab (PDR001), in Patients with Advanced Non-Small Cell Lung Cancer. Clin Cancer Res. 2022 Jun 1;28(11):2313-2320. doi: 10.1158/1078-0432.CCR-21-2742. PMID 35254415
- See also: Randomized, Double Blind, Placebo Controlled "first in-human" Study to Assess the Safety and Tolerability of Single Ascending Oral Doses of PBF-509 in Male Healthy Volunteers" — http://clinicaltrials.gov/ct2/show/NCT01691924?term=pbf-509&rank=1
- See also: Randomized, double blind, placebo controlled, parallel groups study to assess the safety, tolerability and pharmacokinetic profile of PBF-509 (80 mg, 160 mg and 240 mg) after multiple oral doses" in healthy volunteers" — http://clinicaltrials.gov/ct2/show/NCT02111330?term=pbf-509&rank=2